CLINICAL TRIAL: NCT05588141
Title: A Phase I/II Study of Zotiraciclib for Recurrent Malignant Gliomas With Isocitrate Dehydrogenase 1 or 2 (IDH1 or IDH2) Mutations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000860; 000860-C
Record Dates: First submitted 2022-10-15; First posted 2022-10-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01-08

CONDITIONS: Brain Tumor; Cancer
Keywords: Brain Tumor; Glioma; Idh Mutation; Recurrent Disease
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Glioma; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): Escalation/de-escalation dose levels of zotiraciclib given in 28 day cycles
  Interventions: Drug: Zotiraciclib
- 2 (Experimental): Estimated RP2D of zotiraciclib given in 28 day cycles
  Interventions: Drug: Zotiraciclib
- 3 (Experimental): One RP2D dose of zotiraciclib given on the day prior to brain tumor biopsy or resection, a continuation of treatment with estimated RP2D of zotiraciclib given in 28 days cycles following the recovery of the surgery
  Interventions: Drug: Zotiraciclib

INTERVENTIONS:
Drug: Zotiraciclib — Zotiraciclib will be given orally at the DL1, DL-1, or DL 2 once a day on days 1, 4, 8, 11, 15, 18 of every 28-days cycle (18 cycles total).

SUMMARY:
Background:

Diffuse gliomas are tumors that affect the brain and spinal cord. Gliomas that develop in people with certain gene mutations (IDH1 or IDH2) are especially aggressive. Better treatments are needed.

Objective:

To see if a study drug (zotiraciclib) is effective in people with recurrent diffuse gliomas who have IDH1 or IDH2 mutations.

Eligibility:

People aged 15 years and older with diffuse gliomas that returned after treatment. They must also have mutations in the IDH1 or IDH2 genes.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests. They will have tests of their heart function. They will have an MRI of their brain. A new biopsy may be needed if previous results are not available.

Zotiraciclib is a capsule taken by mouth with a glass of water. Participants will take the drug at home on days 1, 4, 8, 11, 15, and 18 of a 28-day cycle. They may also be given medications to prevent side effects of the study drug. The schedule for taking the study drug may vary for participants who will undergo surgery.

Participants will be given a medication diary for each cycle. They will write down the date and time of each dose of the study drug.

Participants will visit the clinic about once a month. They will have a physical exam, blood tests, and tests to evaluate their heart function. An MRI of the brain will be repeated every 8 weeks.

Participants may remain in the study for up to 18 cycles (1.5 years).

DETAILED DESCRIPTION:
Background:

* Zotiraciclib is a multi-kinase inhibitor that has been shown to have anti-glioma effects through transcriptional suppression, mitochondrial dysfunction, and adenosine 5'-triphosphate (ATP) reduction in glioblastoma in our preclinical studies
* Zotiraciclib is orally administered and likely penetrates the blood brain barrier (BBB). There has been a clinical experience in using zotiraciclib as a single agent and in combination with other chemotherapy agents in cancers, including malignant gliomas
* Our phase I study of zotiraciclib and temozolomide (TMZ) in recurrent high-grade astrocytomas determined the maximum tolerated dose (MTD) of zotiraciclib in combination with TMZ and demonstrated the safety of the treatment in recurrent high-grade glioma patients
* Preliminary efficacy analysis of Phase I demonstrated an improved response to zotiraciclib in combination with TMZ in IDH-mutant gliomas compared to the IDH-wildtype counterpart
* A selective vulnerability to zotiraciclib as a single agent was demonstrated in the preclinical models of IDH-mutant gliomas

Objectives:

* Phase I: To estimate recommended phase II dose (RP2D) of zotiraciclib
* Phase II: To determine 12-months progression free survival (PFS) in participants with recurrent glioma, IDH1/2-mutant, World Health Organization (WHO) grade 3 treated with zotiraciclib in comparison with the established brain tumor database matched for tumor molecular characteristics and clinical prognostic factors

Eligibility:

* Age >=15; Karnofsky performance status (KPS) >=70%
* Histological confirmation of diffuse glioma, WHO grades 2-4 with IDH1/2 mutation status confirmed by DNA sequencing
* Have recurrent disease
* Have prior treatment of radiation and/or conventional chemotherapies
* No prior use of bevacizumab as a treatment for a brain tumor

Design:

* This is a phase I/II study to evaluate the safety and efficacy of zotiraciclib as a single agent in recurrent IDH-mutant gliomas.
* Initially, 9-24 participants (Cohort 1) will be assigned to Phase I to estimate recommended phase 2 dose (RP2D) of zotiraciclib.
* Once RP2D is estimated, we will start enrollment into cohorts for Phase II, non-surgical participants (Cohorts 2-4), and surgical (Cohort 5). This trial plans to enroll up 64 evaluable participants.
* Drug will be administered on days 1, 4, 8, 11, 15, 18 in cycles of 28 days for a maximum of 18 cycles. Starting dose is 200 mg. In the case that 200 mg is not tolerable, a lower dose 150 mg, will be evaluated. If 200 mg is tolerated well, a higher dose level will be evaluated at 250 mg.
* Participants in the surgical cohort will get an additional single pre-treatment with one dose of study drug at the RP2D on Day 1 of Cycle 0, followed by brain tumor biopsy or surgical resection within 24 hours on Day 2 of Cycle 0. Approximately 2-4 weeks after surgery or biopsy participants in this Cohort will continue treatment with the study drug and start Day 1 of Cycle 1.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have diffuse glioma, WHO grades 2-4, histologically confirmed by Laboratory of Pathology, NCI.
* IDH1 or IDH2 mutation status confirmed by TruSight(TM) Oncology 500 performed in LP, NCI or prior documentation of IDH1 or IDH2 mutation status
* Participants must have received prior treatment (e.g., radiation, conventional chemotherapy, or vorasidenib) prior to disease progression.
* Participants must have recurrent disease, proven histologically or by imaging studies
* Participants who have undergone prior surgical resection are eligible for enrollment to cohorts 1-4.
* Age >15 years
* Karnofsky >70%
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes >=3,000/microliter
  * absolute neutrophil count (ANC) >=1,500/microliter
  * platelets >100,000/microliter
  * total bilirubin <=2x ULN (ULN 1.3 mg/dl) except for participants with Gilbert Syndrome
  * AST < 3x ULN (ULN 34U/L)
  * ALT < 3x ULN (ULN 55U/L)
  * serum creatinine < 1.5 mg/dL
  * calculated creatinine clearance by CKD-EPI equation > 60 cc/min
* Participants must have recovered from the adverse effects of prior therapy to grade 2 or less (per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0)
* Individuals of child-bearing potential (IOCBP) and men must agree to use highly effective contraception (hormonal, intrauterine device (IUD), abstinence, tube ligation, partner has had a previous vasectomy) at the study entry, for the duration of study treatment, and up to 3 months after the last dose of zotiraciclib
* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 3 months after study treatment discontinuation
* Participants must be scheduled for brain tumor biopsy or surgical resection at NIH (Cohort 5 only)
* The ability of a participant, parent or legal guardian of minor participant to understand and the willingness to sign a written informed consent document. No Legally Authorized Representative can provide initial consent.

EXCLUSION CRITERIA:

* More than one disease relapse in those with initial diagnosis of WHO grade 3-4, or more than two disease relapses in those with initial diagnosis of WHO grade 2 for Phase II. For Phase I enrollment, there are no limits on the number of prior recurrences.
* Prior therapy with:

  * any investigational agent (including IDH mutant inhibitor) and/or standard of care cytotoxic therapy within 28 days prior to treatment initiation
  * vincristine within 14 days prior to treatment initiation
  * nitrosoureas within 42 days prior to treatment initiation
  * procarbazine within 21 days prior to treatment initiation
  * non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, within 7 days prior to treatment initiation
  * surgery within 14 days prior to treatment initiation
  * radiation therapy within 30 days prior to treatment initiation
  * bevacizumab for tumor treatment. Note: participants who received bevacizumab for symptom management, including but not limited to cerebral edema, or pseudo progression can be enrolled
* Prolonged QTc >470ms as calculated by correction formula on screening electrocardiogram (ECG) (QTCf can be used; QTCb can be used for participants with sinus bradycardia)
* Prior invasive malignancies within the past 3 years prior to study treatment initiation (with the exception of non-melanoma skin cancers, carcinoma in situ of the cervix, melanoma in situ, or any localized cancer for whom the systemic standard of care therapy is not required)
* History of allergic reactions attributed to compounds of similar chemical composition to zotiraciclib, such as flavopiridol
* Pregnancy (confirmed with beta-HCG serum or urine pregnancy test performed at screening)
* Uncontrolled intercurrent illness or social situations that would limit compliance with study requirements
* Uncontrolled primary diabetes mellitus

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2032-08-02 (Estimated)

PRIMARY OUTCOMES:
To determine 12 months PFS in participants w/ recurrent glioma, IDH1/2-mutant, WHO grade 3 treated w/ zotiraciclib in comparison w/ the established brain tumor database matched for tumor molecular characteristics and clinical prognostic factors | 12 Months
  Proportion of patients that have progressive disease after 12 months
To estimate recommended phase II dose (RP2D) of zotiraciclib | 28 days
  Number of DLTs within the DLT Period

SECONDARY OUTCOMES:
To determine the efficacy of treatment with zotiraciclib in participants with recurrent glioma, IDH1/2-mutant WHO grade 3 in comparison with the established brain tumor database by 3 years PFS rate | 3 years
  Amount of time until disease progression from initiation of study therapy as compared with data of the brain tumor database
To determine the safety of zotiraciclib in participants with recurrent glioma, IDH1/2-mutant WHO grades 2-4 | Day 1 of Cycle 0 (Cohort 5) or Day 1 of Cycle 1 (Cohorts 1-4) through 30 days after the study agent was last administered will be collected on the days study drug is administered, and at the safety follow up visit.
  Type, grade and frequency of adverse events
To determine the efficacy of treatment with zotiraciclib in participants with recurrent glioma, IDH1/2-mutant WHO grade 3 in comparison with the established brain tumor database by 5 years overall survival (OS) rate | 5 years
  Amount of time subject survives after initiation of study therapy as compared with data of the brain tumor database

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Yuan Y, Hess KR, Hilsenbeck SG, Gilbert MR. Bayesian Optimal Interval Design: A Simple and Well-Performing Design for Phase I Oncology Trials. Clin Cancer Res. 2016 Sep 1;22(17):4291-301. doi: 10.1158/1078-0432.CCR-16-0592. Epub 2016 Jul 12. PMID 27407096
- [Background] Miller JJ, Loebel F, Juratli TA, Tummala SS, Williams EA, Batchelor TT, Arrillaga-Romany I, Cahill DP. Accelerated progression of IDH mutant glioma after first recurrence. Neuro Oncol. 2019 May 6;21(5):669-677. doi: 10.1093/neuonc/noz016. PMID 30668823
- [Background] Wu J, Yuan Y, Long Priel DA, Fink D, Peer CJ, Sissung TM, Su YT, Pang Y, Yu G, Butler MK, Mendoza TR, Vera E, Ahmad S, Bryla C, Lindsley M, Grajkowska E, Mentges K, Boris L, Antony R, Garren N, Siegel C, Lollo N, Cordova C, Aboud O, Theeler BJ, Burton EM, Penas-Prado M, Leeper H, Gonzales J, Armstrong TS, Calvo KR, Figg WD, Kuhns DB, Gallin JI, Gilbert MR. Phase I Study of Zotiraciclib in Combination with Temozolomide for Patients with Recurrent High-grade Astrocytomas. Clin Cancer Res. 2021 Jun 15;27(12):3298-3306. doi: 10.1158/1078-0432.CCR-20-4730. Epub 2021 Mar 30. PMID 33785481
- [Derived] Pang Y, Li Q, Sergi Z, Yu G, Kim O, Lu P, Chan M, Sang X, Wang H, Ranjan A, Robey RW, Soheilian F, Tran B, Nunez FJ, Zhang M, Song H, Zhang W, Davis D, Gilbert MR, Gottesman MM, Liu Z, Thomas CJ, Castro MG, Gujral TS, Wu J. Exploiting the therapeutic vulnerability of IDH-mutant gliomas with zotiraciclib. iScience. 2025 Mar 25;28(4):112283. doi: 10.1016/j.isci.2025.112283. eCollection 2025 Apr 18. PMID 40241769
- [Derived] Pang Y, Li Q, Sergi Z, Yu G, Sang X, Kim O, Wang H, Ranjan A, Merchant M, Oudit B, Robey RW, Soheilian F, Tran B, Nunez FJ, Zhang M, Song H, Zhang W, Davis D, Gilbert MR, Gottesman MM, Liu Z, Khan J, Thomas CJ, Castro MG, Gujral TS, Wu J. Exploiting the therapeutic vulnerability of IDH-mutant gliomas with zotiraciclib. bioRxiv [Preprint]. 2024 Jan 2:2023.06.29.547143. doi: 10.1101/2023.06.29.547143. PMID 37786680
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000860-C.html